CLINICAL TRIAL: NCT05725096
Title: Role of the Screening with Coronary Computed Tomography Angiography on Lipid Management and Risk Factors Control in an Asymptomatic Chinese Population: a Community-based, Prospective Randomised Trial
Brief Title: Role of Coronary CTA on Lipid Management and Risk Factors Control in an Asymptomatic Chinese Population
Acronym: RESPECT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang longjiang,MD (Other)
Responsible Party: Sponsor-Investigator, Zhang longjiang,MD, Principal Investigator : Zhang longjiang, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022DZKY-056-01
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Statin; Cardiovascular Risk Factors; Primary Prevention; Adherence, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCTA-based strategy group (Active Comparator): Subjects will be managed following the CCTA -based coronary heart disease prevention strategy for lipid-lowering treatment and follow-up.
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography
- Chinese guidelines for lipid management (2023) (Sham Comparator): The baseline assessment will be completed on the same day as consent is gained. Every subjects will complete a comprehensive assessment including questionnaires and objective assessments.
  Interventions: Other: Traditional cardiovascular risk stratification

INTERVENTIONS:
Diagnostic Test: Coronary Computed Tomography Angiography — Intervention strategies according to CCTA results
  Arms: CCTA-based strategy group
Other: Traditional cardiovascular risk stratification — Intervention strategies according to traditional cardiovascular risk stratification based on Chinese guidelines for lipid management (2023)
  Arms: Chinese guidelines for lipid management (2023)

SUMMARY:
The primary objective of this study is to determine whether coronary computed tomography angiography (CCTA) -based coronary heart disease(CHD) prevention strategy improves lipid-lowering treatment and cardiovascular risk factor control compared with traditional CHD prevention strategy, guided by a cardiovascular risk score.

DETAILED DESCRIPTION:
At present, doctors usually use a "risk score" to identify people at risk of heart disease who may benefit from medical treatment. In the RESPECT study the investigator will compare this "risk score" to coronary CTA scan. In this study the investigator would like to determine the effect of coronary CTA scan on lipid-lowering treatment and cardiovascular risk factor control.

This study will recruit 3400 eligible community volunteers (asymptomatic individuals free of any known cardiovascular event) aged 40 to 69 years, then, randomized (1:1) them to receive individualized primary prevention programs for coronary heart disease based on CCTA results or traditional risk score, as recommended in the Chinese CVD prevention guidelines. The intervention strategies in this study are consistent with RESPECT trial.

The investigator will assess the difference of lipid-lowering treatment and cardiovascular risk factor control between two groups 12 months later. Furthermore, the investigator will present the results of subclinical coronary atherosclerosis in participants who have undergone coronary CTA scans. This will help us understand the prevalence of subclinical coronary atherosclerotic disease in an asymptomatic Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Nanjing residents who have no plans to leave in the next 5 years
2. Aged from 40 to 69 years
3. Free of any known clinically cardiovascular disease Able to comprehend and sign an informed consent form

Exclusion Criteria:

1. Serious liver dysfunction, defined as AST or ALT > 3 times the normal upper limit
2. Chronic kidney disease (CKD) > stage 4, defined as eGFR < 30 ml/min/1.73 m2
3. Prior CCTA or invasive coronary angiography within the last 5 years
4. Any contraindications for CCTA
5. Previous use of statin or non-statin lipid-lowering medication (such as ezetimibe, PCSK9 inhibitor and XueZhiKang)
6. Life expectancy < 3 years
7. Other reasons the researcher deems inappropriate to attend

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants taking lipid-lowering medication regularly at both 6 and 12 months | 12 months
  Taking lipid-lowering medication regularly defined as taking the established lipid-lowering medication (including statin, ezetimibe, xuezhikang and PCSK9 inhibitor) at least 24 days during the past 30 days.

SECONDARY OUTCOMES:
The proportion of participants achieving LDL-C targets at 12 months | 12 months
  The LDL-C treatment goals are made according to Chinese guideline
The proportion of participants taking lipid-lowering medication regularly at 12 months. | 12 months
  The proportion of participants taking lipid-lowering medication regularly at 12 months. Taking lipid-lowering medication regularly defined as taking the established lipid-lowering medication (including statin, ezetimibe, xuezhikang and PCSK9 inhibitor) at least 24 days during the past 30 days.
Cardiovascular events | 12 months
  Number of participants diagnosed with coronary heart disease, stroke (hemorrhagic and ischemic), TIA or cardiovascular death
Prevalence of subclinical coronary atherosclerotic disease | baseline
  Proportion of subjects with coronary atherosclerosis in participants who underwent coronary CTA scan (%)
LDL-C levels | 12 months
  Compare the difference in LDL-C concentration between baseline and one year later, with the measurement unit being mmol/L.
Hypertension control | 12 months
  SBP<140mmHg and DBP<90mmHg
Diabetic control | 12 months
  HbA1c <53 mmol/mol (7.0%)
Smoking cessation | 12 months
  Proportion of subjects who changed smoking habits (%)
Exercise | 12 months
  Change in activity levels measured through international physical activity questionnaire
Quality of life/Anxiety and Depression | 12 months
  Change in quality of life measured through PHQ-9 (patient health questionnaire): anxiety and depression score (%)

OTHER OUTCOMES:
Changes in renal function before and after CCTA examination | All participants in the experimental group completed CCTA 1 month later
  The status of kidney function is represented by eGFR.

CONTACTS AND LOCATIONS:
Overall Officials: Trail Manager, Study Chair — Jinling Hospital,Nanjing University School of Medicine,Nanjing,China
Locations (1):
- Research Institute Of Medical Imaging Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Guo X, Li J, Zhu Y, Li Y, Jiang J, Zuo R, Xu W, Ma J, Li C, Yang J, Liu Y, Zhao M, Tian D, Wang X, Sun J, Wu B, Wang C, Jiang P, Zhang J, Zhong J, Zhou C, Yi D, Bao X, Cai J, Chen Y, Cheng X, Gong H, Wei Y, Liu Y, Zhang LJ. Role of the screening with coronary computed tomography angiography on lipid management and risk factors control in an asymptomatic Chinese population: a community-based, parallel-group, open-label, randomized clinical trial (RESPECT2). Trials. 2024 Sep 30;25(1):635. doi: 10.1186/s13063-024-08469-z. PMID 39350195